CLINICAL TRIAL: NCT00716131
Title: ALS Tissue Donation Program
Brief Title: Amyotrophic Lateral Sclerosis (ALS) Tissue Donation Program
Status: Completed | Type: Observational
Sponsor: Drexel University College of Medicine (Other)
Collaborators: MDA/ALS Center of Hope (Other)
Responsible Party: Principal Investigator, Christine Barr, Research Nurse Coordinator, Drexel University
Organization: Drexel University (Other)
Other Study IDs: Internal-16827
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Amyotrophic Lateral Sclerosis; Neurodegenerative Disease; Motor Neuron Disease
Keywords: Amyotrophic Lateral Sclerosis; Cerebrospinal Fluid; Neurodegenerative Disease; Motor Neuron Disease; Autonomic Nervous System; Neurodegenerative Diseases; Movement Disorders
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases; Motor Neuron Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood (Serum and DNA) Urine (Serum and DNA) CSF Blood specimens and tissue specimens (from brain, spinal cord, gastrointestinal tract, skeletal muscle and peripheral nerve)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- ALS: Diagnosed with ALS or other motor system disorder including PLS, Bulbar Palsy or Motor neuropathy
- Neuro: Diagnosed with other chronic neurologic illnesses (Alzheimers, multiple sclerosis, migraines, etc)
- Healthy: Normal Controls
- Autopsy

SUMMARY:
Despite significant progress in the identification of mechanisms involved in motor neuron degeneration in Amyotrophic Lateral Sclerosis (ALS) and other motor system diseases, the actual pathogenesis and cause of these diseases remains unknown. Effective treatment of these diseases are dependent on the elucidation of their causes. The availability of diseased and control human tissues will be a critical resource for this research progress. . Samples of serum, spinal fluid, and urine from patients with motor system diseases can be used to study biochemical and genetic differences compared to tissues of neurologic disease controls and normal controls. Furthermore, the availability of autopsied CNS, PNS, as well as other tissues from patients with ALS or suspected ALS are useful for current and future research studies into the disease. Therefore, we propose to institute a Tissue Bank containing blood, urine, and cerebrospinal fluid donated from not only ALS and other motor neuron disease patients, but also those with other neurologic diseases and normals whose tissue can be used as controls. In addition there will be an autopsy band for post-mortem specimens of ALS and other motor neuron disease patients. Each specimen, whether from a living patient or autopsy will be de-identified and accompanied by a standard set of clinical information collected from the medical records in order that each specimen is characterized with the relevant clinical information to maximize the usefulness of the specimens.

Once established, this tissue bank will provide a resource in which a large number of samples will be readily available and expedite research by circumventing the delays in collecting specimens prospectively. These specimens will be used for research in the ALS Center of Hope at Drexel University College of Medicine and shared with any outside investigator with a valid IRB approved protocol.

DETAILED DESCRIPTION:
Despite significant progress in the identification of mechanisms involved in motor neuron degeneration in Amyotrophic Lateral Sclerosis (ALS) and other motor system diseases, the actual pathogenesis and cause of these diseases remains unknown. Effective treatment of these diseases are dependent on the elucidation of their causes. The availability of diseased and control human tissues will be a critical resource for this research progress. . Samples of serum, spinal fluid, and urine from patients with motor system diseases can be used to study biochemical and genetic differences compared to tissues of neurologic disease controls and normal controls. Furthermore, the availability of autopsied CNS, PNS, as well as other tissues from patients with ALS or suspected ALS are useful for current and future research studies into the disease. Therefore, we propose to institute a Tissue Bank containing blood, urine, and cerebrospinal fluid donated from not only ALS and other motor neuron disease patients, but also those with other neurologic diseases and normals whose tissue can be used as controls. In addition there will be an autopsy band for post-mortem specimens of ALS and other motor neuron disease patients. Each specimen, whether from a living patient or autopsy will be de-identified and accompanied by a standard set of clinical information collected from the medical records in order that each specimen is characterized with the relevant clinical information to maximize the usefulness of the specimens.

Once established, this tissue bank will provide a resource in which a large number of samples will be readily available and expedite research by circumventing the delays in collecting specimens prospectively. These specimens will be used for research in the ALS Center of Hope at Drexel University College of Medicine and shared with any outside investigator with a valid IRB approved protocol.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ALS or other motor system disorder including PLS, Bulbar Palsy or Motor neuropathy
* Diagnosed with other chronic neurologic illnesses (Alzheimers, multiple sclerosis, migraines, etc)
* Normal Controls
* In the case of spinal fluid collection, the patient will be undergoing a diagnostic lumbar puncture as part of the work-up

Exclusion Criteria:

* Any person with a non-neurologic chronic and poorly controlled systemic illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALS clinic patients at MDA/ALS Center of Hope, along with families and caregivers. Also those with ALS who have donated their bodies to research.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2007-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
None Specified | None Specified
  No primary outcome measure is specified for this study. Purpose of the study is to collect deidentified biological specimens which will be used to expedite other IRB approved studies.

CONTACTS AND LOCATIONS:
Overall Officials: Terry D Heiman-Patterson, MD, Principal Investigator — Drexel University College of Medicine
Locations (1):
- MDA/ALS Center of Hope, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The purpose of this protocol is to collect and bank tissue specimens.